CLINICAL TRIAL: NCT02494752
Title: Potential of Mesenchymal Stem Cell Enriched Adipose Tissue Grafting for Contour Deformities of Face
Brief Title: Role of Mesenchymal Stem Cells in Fat Grafting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King Edward Medical University (Other)
Responsible Party: Principal Investigator, Muhammad Mustehsan Bashir, Associate professor of Plastic Surgery, King Edward Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 229/RC/KEMU
Record Dates: First submitted 2015-07-04; First posted 2015-07-10 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-07

CONDITIONS: Romberg's Disease; Craniofacial Microsomia; Lipodystrophy; Mixed Connective Tissue Disease
Keywords: Contour deformities of face; autologous fat grafting; Post traumatic facial contour defects
MeSH Terms: conditions — Facial Hemiatrophy; Goldenhar Syndrome; Lipodystrophy; Mixed Connective Tissue Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stem cell enriched (Experimental): Fat graft will be enriched with ex vivo expanded stem cells
  Interventions: Procedure: Fat graft enriched with ex vivo expanded stem cells
- Non stem cell enriched (Active Comparator): Fat graft will not be enriched with ex vivo expanded stem cells
  Interventions: Procedure: Fat graft not enriched with ex vivo expanded stem cells

INTERVENTIONS:
Procedure: Fat graft enriched with ex vivo expanded stem cells — Fat graft will be enriched with ex vivo expanded stem cells
  Arms: Stem cell enriched
Procedure: Fat graft not enriched with ex vivo expanded stem cells — Fat graft will not be enriched with ex vivo expanded stem cells
  Arms: Non stem cell enriched

SUMMARY:
Contour deformity of face causes both functional as well as aesthetic problems for the patient. Fat being an autologous tissue source is considered as an ideal soft-tissue filler because it is abundant, readily available, inexpensive, host compatible, and can be harvested easily and repeatedly. However absorption of grafted fat is a major problem resulting in lack of consistency of final clinical outcome. Adipose tissue derived mesenchymal stem cells have the potential to enhance the viability of the grafted fat and the reliability of the final outcome of surgery. In the current study potential of mesenchymal stem cells will be studied by comparing two groups of patients requiring fat grafting for contour deformities of face. Control group will have fat graft with out enrichment with stem cells whereas experimental group will have their fat graft enriched with mesenchymal stem cells. Comparison will be made regarding viability of grafted fat in two groups.

DETAILED DESCRIPTION:
Contour deformities of the face requiring soft tissue augmentation often result from conditions such as congenital disorders, acquired diseases, and traumatic and developmental deformities. Significant contour deformity of face causes both functional as well as aesthetic problems for the patient. Conventionally, these problems are treated by allogenic fillers, major flap surgery and fat grafting.1 However; different problems are associated with above mentioned treatment options. For example, allogenic fillers are foreign material that poses not only allergic reactions but also rapid absorption at the site of application. Similarly, flap surgery, in the form of pedicled and free flaps, produces considerable donor site morbidity. In addition, fine- tuning is impossible with flap, and tissue transferred in the form of flap may act as blob.

Autologous fat grafting has gained pervasive acceptance for the management of contour deformities of the face. Fat being an autologous tissue source is considered as an ideal soft-tissue filler because it is abundant, readily available, inexpensive, host compatible, and can be harvested easily and repeatedly.2 Although the practice of fat grafting is not new and it is a safe and natural method of soft-tissue augmentation, the viability and reliability of transplanted fat grafts remains poorly studied. One major concern is the lack of consistency of final clinical outcome, which often requires multiple fat grafting procedures making it expensive. Rate of fat absorption may reach up to 40% to 80%.However, previously published data have failed to produce a cohesive algorithm of the required components for successful, consistent and durable fat transplantation.3 In order to overcome problems associated with fat grafting, other innovative techniques are required.

The role of fat auto-transplantation in plastic surgery has evolved from a controversial technique designed for simple volume augmentation to the foundation for the innovative and burgeoning field of regenerative medicine. This is based on the fact that adipose tissue contains adipocytes and the stromal vascular fraction (SVF) consisting of multiple cell types such as circulating blood cells, fibroblasts, pericytes, endothelial cells, and mesenchymal stem cells (MSCs). Adipocytes account for 20 percent or fewer of the total number of cells in adipose tissue4whereasthere are only 3% MSCs in SVF of adipose tissue.5 Although this percentage is relatively low, this cell type is the main contributor in overall healing process. MSCs derived from adipose tissue (AT-MSCs) have high proliferative potential and ability to differentiate into mesenchymal (adipose, bone, cartilage) and non-mesenchymal (neuron like cells) lineages.6,7,8 AT-MSCs have been shown to enhance angiogenesis, decrease apoptosis and modify the local inflammatory response owing to their immunosuppressive and immunomodulatory properties.9 Therefore, the current study is designed to evaluate the effect of fat grafting and AT-MSCs together on contour deformities of face. By combining traditional fat graft with AT-MSCs, tissue viability and therefore the consistency of graft survival may be improved. In the current model investigators propose that transferred fat may act as a natural scaffold and temporary filler to restore the volume immediately while AT-MSCs will start participating in multiple parameters of tissue regeneration. This model supports the "host replacement theory" that has been put forward to describe how fat grafts survive after they are transplanted.10 Due to problems associated with fat grafting alone, it is desirable to solve such issues by using innovating techniques. In the current study investigators propose the novel idea of enrichment of conventional fat graft with ex-vivo expanded AT-MSCs to enhance the viability of the grafted fat and the reliability of the final outcome of surgery. Recent animal studies have suggested that AT-MSCs that have been expanded before administration could help preserve grafted fat and improve outcomes.11 Thus rationale of current study is to compare the outcome of conventional fat grafting with stem cell enriched fat grafting for contour deformities of face. If enrichment of fat graft with AT-MSCs can decrease its absorption rate, this innovative strategy can make fat transfer a reliable option for soft tissue augmentation. This can definitely improve final clinical outcome at lesser cost and reduced donor site morbidity

ELIGIBILITY:
Inclusion Criteria:

* Patients with congenital and acquired contour deformities of face requiring soft tissue augmentation .
* Must be 16-60 years of age
* Must be American Society of Anesthesiology (ASA) class 1 and 2

Exclusion Criteria:

* Patients with contour deformities in which skin is adherent to facial skeleton
* Contour deformities underlying skin grafted areas of face
* Abdominal skin pinch thickness less than 3 inch

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in thickness of subcutaneous tissue | 24 weeks
  Objective assessment will be made by doing baseline B mode colour Doppler ultrasonography of the treated area.The operator blinded to the group allocation will measure the thickness of the subcutaneous tissue (in millimeters) in the treated area during the baseline examination with ultrasound B-mode. In order to have a reproducible measurement in subsequent examinations, the operator will look for and note down precise anatomical landmarks or, in case of large areas, will mark the points with an indelible marker, saving a digital image for future reference. Patients will again under go ultrasonography of the treated area at 24 weeks post treatment. During this repeat ultra sonography same operator will again measure the subcutaneous thickness of the treated in millimeters. The difference in two measurements will be noted down as residual volume. Means of residual volumes in two groups will be compared.

SECONDARY OUTCOMES:
Change from base line in post operative appearance | 24 weeks
  Subjective assessment will be done by taking photographs preoperatively and 24 weeks post treatment months under standard conditions of light, distance, views and camera make. Two plastic surgeons blinded to group allocation will rate post operative appearance as satisfactory/unsatisfactory by comparing pre and post operative photographs.

REFERENCES:
- [Background] Cheong YW, Lo LJ. Facial asymmetry: etiology, evaluation, and management. Chang Gung Med J. 2011 Jul-Aug;34(4):341-51. PMID 21880188
- [Background] Bucky LP, Kanchwala SK. The role of autologous fat and alternative fillers in the aging face. Plast Reconstr Surg. 2007 Nov;120(6 Suppl):89S-97S. doi: 10.1097/01.prs.0000248866.57638.40. PMID 18090347
- [Background] Gir P, Brown SA, Oni G, Kashefi N, Mojallal A, Rohrich RJ. Fat grafting: evidence-based review on autologous fat harvesting, processing, reinjection, and storage. Plast Reconstr Surg. 2012 Jul;130(1):249-258. doi: 10.1097/PRS.0b013e318254b4d3. PMID 22743888
- [Background] Brown SA, Levi B, Lequex C, Wong VW, Mojallal A, Longaker MT. Basic science review on adipose tissue for clinicians. Plast Reconstr Surg. 2010 Dec;126(6):1936-1946. doi: 10.1097/PRS.0b013e3181f44790. PMID 21124133
- [Background] Baer PC, Geiger H. Adipose-derived mesenchymal stromal/stem cells: tissue localization, characterization, and heterogeneity. Stem Cells Int. 2012;2012:812693. doi: 10.1155/2012/812693. Epub 2012 Apr 12. PMID 22577397
- [Background] Choudhery MS, Badowski M, Muise A, Pierce J, Harris DT. Donor age negatively impacts adipose tissue-derived mesenchymal stem cell expansion and differentiation. J Transl Med. 2014 Jan 7;12:8. doi: 10.1186/1479-5876-12-8. PMID 24397850
- [Background] Choudhery MS, Badowski M, Muise A, Harris DT. Comparison of human mesenchymal stem cells derived from adipose and cord tissue. Cytotherapy. 2013 Mar;15(3):330-43. doi: 10.1016/j.jcyt.2012.11.010. Epub 2013 Jan 11. PMID 23318344
- [Background] Choudhery MS, Badowski M, Muise A, Pierce J, Harris DT. Cryopreservation of whole adipose tissue for future use in regenerative medicine. J Surg Res. 2014 Mar;187(1):24-35. doi: 10.1016/j.jss.2013.09.027. Epub 2013 Oct 8. PMID 24268882
- [Background] Tiryaki T, Findikli N, Tiryaki D. Staged stem cell-enriched tissue (SET) injections for soft tissue augmentation in hostile recipient areas: a preliminary report. Aesthetic Plast Surg. 2011 Dec;35(6):965-71. doi: 10.1007/s00266-011-9716-x. Epub 2011 Apr 13. PMID 21487913
- [Background] Eto H, Kato H, Suga H, Aoi N, Doi K, Kuno S, Yoshimura K. The fate of adipocytes after nonvascularized fat grafting: evidence of early death and replacement of adipocytes. Plast Reconstr Surg. 2012 May;129(5):1081-1092. doi: 10.1097/PRS.0b013e31824a2b19. PMID 22261562
- [Background] Gir P, Oni G, Brown SA, Mojallal A, Rohrich RJ. Human adipose stem cells: current clinical applications. Plast Reconstr Surg. 2012 Jun;129(6):1277-1290. doi: 10.1097/PRS.0b013e31824ecae6. PMID 22634645
- [Background] Kolle SF, Fischer-Nielsen A, Mathiasen AB, Elberg JJ, Oliveri RS, Glovinski PV, Kastrup J, Kirchhoff M, Rasmussen BS, Talman ML, Thomsen C, Dickmeiss E, Drzewiecki KT. Enrichment of autologous fat grafts with ex-vivo expanded adipose tissue-derived stem cells for graft survival: a randomised placebo-controlled trial. Lancet. 2013 Sep 28;382(9898):1113-20. doi: 10.1016/S0140-6736(13)61410-5. PMID 24075051
- [Background] Bollero D, Pozza S, Gangemi EN, De Marchi A, Ganem J, A M el K, Faletti C, Stella M. Contrast-enhanced ultrasonography evaluation after autologous fat grafting in scar revision. G Chir. 2014 Nov-Dec;35(11-12):266-73. PMID 25644727
- [Derived] Bashir MM, Sohail M, Ahmad FJ, Choudhery MS. Preenrichment with Adipose Tissue-Derived Stem Cells Improves Fat Graft Retention in Patients with Contour Deformities of the Face. Stem Cells Int. 2019 Nov 20;2019:5146594. doi: 10.1155/2019/5146594. eCollection 2019. PMID 31827528